CLINICAL TRIAL: NCT03893877
Title: Noninvasive Mechanic Ventilation With Nasal Mask is Better Than Oxygen Delivery Via Nasal Cannula for Dental Treatments in Children Performed Under Deep Sedation: Randomised ,Prospective, Clinical Study
Brief Title: Comparison of Oxygenation Methods in Sedation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, seher orbay yasli, assistant professor, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/475
Record Dates: First submitted 2018-11-06; First posted 2019-03-28 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Deep Sedation
MeSH Terms: interventions — Cannula

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal cannula (Experimental): device:nasal cannula will be applied to patients for oxygenation under deep sedation
  Interventions: Device: nasal cannula
- nasal mask (Active Comparator): device:nasal mask will be applied to patients for oxygenation under deep sedation
  Interventions: Device: nasal mask

INTERVENTIONS:
Device: nasal cannula — experimental group will be applied nasal cannula
  Arms: nasal cannula
Device: nasal mask — active comparator group will be applied nasal mask
  Arms: nasal mask

SUMMARY:
Abstract

Backgrounds and objectives:

Dental treatments, especially in children who can not be cooperated, may require deep sedation due to intense anxiety and fear. During sedation oxygen is usually given to the patients by nasal cannula. Investigators want to use nasal mask for non-invasive mechanical ventilation for oxygenation of the patient during sedation for dental treatment and described it with nasal cannula.

Methods:

Seventy three children classified as ASA 1 or 2, aged between 3 to 17 will be included for this study. During deep sedation procedure group M will be applied nasal mask in order to noninvazive mechanical ventilation, group C will be applied nasal cannula connected to the oxygen flowmeter.

DETAILED DESCRIPTION:
Majority of dental treatments can be performed under local anesthesia. However, this is not always possible for pediatric non-cooperative patients with severe anxiety. In these cases, unpleasant dental experiences may lead to dental phobia when they become adults. For such patients requiring short-term dental procedures, sedation can best choice.

In sedative procedures of patients it is necessary to delivery oxygen to the patient's respiratory system. This can achieved by means of nasal cannulas or interface masks like nasal mask which are connected to the oxygen flowmeter of the anesthesia machine. Investigators hypotezed that oxygen delivery via non-invazive machanic ventilation with nasal mask which is connected to the anesthesia-breathing circuit unit could be better than nasal cannula connected to the oxygen flowmeter of the anesthesia machine during deep sedation for dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients aged betweeen 3-17
* patients with wn ASA( American Society of Anesthesiologists) score 1-2

Exclusion Criteria:

* patients under 3 years old
* patients above of ASA score 2

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2018-11-04 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
effects of non invasive mechanical ventilation on oxygen saturation during deep-sedated patients. | 30 MINUTES
  In investigators want to discuss the differences of oxygen saturations between nasal cannula and nasal mask.sedative procedures of patients it is necessary to delivery oxygen to the patient's respiratory system. This can achieved by means of nasal cannulas or interface masks like nasal mask which are connected to the oxygen flowmeter of the anesthesia machine.

CONTACTS AND LOCATIONS:
Overall Officials: Seher O Yasli, Principal Investigator — Ercıyes University faculty of dentistry
Locations (1):
- Seher Orbay Yasli, Kayseri, Turkey (Türkiye)